CLINICAL TRIAL: NCT02259179
Title: A Phase 1 Bioequivalence Study of Naltrexone SR/Bupropion SR Combination Trilayer Tablets From Two Manufacturers in Healthy Subjects
Brief Title: Bioequivalence Study Comparing Naltrexone SR/Bupropion SR Trilayer Tablets From Two Manufacturers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Orexigen Therapeutics, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: NB-240
Record Dates: First submitted 2014-10-03; First posted 2014-10-08 (Estimated); Last update posted 2014-12-11 (Estimated); Status verified 2014-12

CONDITIONS: Healthy
Keywords: Obesity; Overweight; Contrave; Antiobesity agents; Antiobesity drugs; Weight loss drug; Bioequivalence; Pharmacokinetic
MeSH Terms: conditions — Obesity; Overweight | interventions — bupropion hydrochloride, naltrexone hydrochoride drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fed Group (Active Comparator): Reference and test product naltrexone SR/bupropion SR combination trilayer tablets tested in the fed state.
  Interventions: Drug: Reference naltrexone 8 mg SR/bupropion 90 mg SR combination trilayer tablets (2 tablets); Drug: Test naltrexone 8 mg SR/bupropion 90 mg SR combination trilayer tablets (2 tablets)
- Fasted group (Active Comparator): Reference and test product naltrexone SR/bupropion SR combination trilayer tablets tested in the fasted state.
  Interventions: Drug: Reference naltrexone 8 mg SR/bupropion 90 mg SR combination trilayer tablets (2 tablets); Drug: Test naltrexone 8 mg SR/bupropion 90 mg SR combination trilayer tablets (2 tablets)

INTERVENTIONS:
Drug: Reference naltrexone 8 mg SR/bupropion 90 mg SR combination trilayer tablets (2 tablets)
  Other Names: Contrave
Drug: Test naltrexone 8 mg SR/bupropion 90 mg SR combination trilayer tablets (2 tablets)

SUMMARY:
This is a Phase 1, open-label, randomized, single-dose, 2-way crossover study in healthy adult subjects to assess the bioequivalence of naltrexone SR/bupropion SR combination trilayer tablets prepared at two different manufacturing sites. The pharmacokinetics of the two drug products will be evaluated separately in the fed and fasted state.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, 18 to 60 years of age, inclusive
2. Be in good general health, without any clinically significant medical history, physical examination findings, or laboratory results at Screening or Day -1
3. Body mass index (BMI) of 18 to 30 kg/m2, inclusive, at Screening

Exclusion Criteria:

1. Acute (within 28 days of Day -1) or chronic illness
2. History (within the last 20 years) of seizures, cranial trauma, bulimia, anorexia nervosa, or other conditions that may predispose the subject to seizures; or previous medical treatment with anticonvulsants of any type
3. History of mania or current diagnosis of active psychosis
4. Acute depressive illness, including new onset of depression or acute exacerbation of symptoms
5. Use of any prescription medication within 14 days prior to Day -1, with the exception of hormonal contraceptive or hormonal replacement therapy (HRT) at a stable dose for at least 28 days prior to Day -1
6. Use of any over-the-counter medications, including dietary/nutritional and herbal supplements, within 24 hours prior to study drug intake on Day 1
7. Use of bupropion- or naltrexone-containing products within 28 days prior to Day -1, or history of hypersensitivity or intolerance to naltrexone or bupropion
8. Have donated blood or have had significant blood loss within 90 days prior to Day -1; or have donated plasma within 7 days prior to Day -1
9. Hemoglobin concentration <11 g/dL at Screening
10. Blood pressure >140/90 mm Hg at Screening or Day -1
11. Women who are pregnant or trying to become pregnant, have a positive pregnancy test at Screening or Day -1, are currently breast-feeding, or are of childbearing potential (including perimenopausal women who have had a menstrual period within 1 year prior to Day -1) and are not willing to practice effective birth control. Women who are surgically sterile (including bilateral tubal ligation, tubal occlusion, hysterectomy or oophorectomy) are not considered to be of childbearing potential.
12. Drug or alcohol abuse or dependence within 6 months prior to Screening, or positive urine drug screen at Screening or Day -1
13. Regular daily use of tobacco products, including inhaled tobacco (e.g., cigarettes, cigars, pipes), chewing tobacco or snuff, or nicotine replacement products (including electronic cigarettes or nicotine vaporizers) within 28 days prior to Day -1
14. Unwilling to refrain from consumption of any citrus products (e.g., whole fruit, juice or products containing orange, grapefruit, or pomelo), alcohol or caffeine/xanthine-containing foods or beverages for 48 hours before study drug intake in each treatment period (Days 1 and 15) until 72 hours postdose (Days 4 and 18)
15. Inability or unwillingness to consume a standardized high-fat breakfast as provided at the study clinic on Days 1 and 15
16. Inability to comply with all required study procedures and schedule, inability to speak and read English, or unwillingness or inability to give written informed consent
17. Employee or immediate family member of the sponsor (or designee) or study site research staff
18. Use of any investigational drug, device, or procedure within 30 days prior to Day -1

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2014-09; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Cmax | 0-96 hours post-dose
  Maximum observed plasma concentration
AUC(0-t) | 0-96 hours post-dose
  Area under the plasma concentration-time curve from 0 hour to the time of the last quantifiable concentration
AUC(0-inf) | 0-96 hours post-dose
  Area under the plasma concentration-time curve from 0 hour extrapolated to infinity

CONTACTS AND LOCATIONS:
Overall Officials: Senior Vice President Head of Global Development, Study Director — Orexigen Therapeutics, Inc
Locations (1):
- Quintiles Phase One Services, LLC, Overland Park, Kansas, United States